CLINICAL TRIAL: NCT02988115
Title: A Randomized, Double-Blind, Parallel Group, Multicenter Study to Evaluate the Efficacy and Safety of Bempedoic Acid (ETC-1002) 180 mg Compared to Placebo Added to Background Lipid-Modifying Therapy in Patients With Elevated LDL-C Who Are Statin Intolerant
Brief Title: Evaluation of the Efficacy and Safety of Bempedoic Acid (ETC-1002) in Patients With Hyperlipidemia and Statin Intolerant
Acronym: CLEAR Serenity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Esperion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1002-046
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Results first posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Hypercholesterolemia; Atherosclerotic Cardiovascular Disease; Statin Adverse Reaction
Keywords: hyperlipidemia; cholesterol; familial hypercholesterolemia; atherosclerotic cardiovascular disease; ASCVD; HeFH; LDL; statin intolerance
MeSH Terms: conditions — Hypercholesterolemia; Atherosclerosis; Hyperlipidemias; Hyperlipoproteinemia Type II | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bempedoic acid (Experimental): bempedoic acid 180 mg tablet taken orally, daily. Patients remain on ongoing lipid-modifying therapy (not study provided)
  Interventions: Drug: bempedoic acid
- placebo (Placebo Comparator): Matching placebo tablet taken orally, daily. Patients remain on ongoing lipid-modifying therapy (not study provided)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: bempedoic acid — bempedoic acid 180 mg tablet
  Other Names: ETC-1002
  Arms: bempedoic acid
Other: placebo — Matching placebo tablet
  Other Names: placebo control
  Arms: placebo

SUMMARY:
The purpose of this study is to determine if bempedoic acid (ETC-1002) is effective and safe versus placebo in patients with elevated LDL cholesterol and who are statin-intolerant.

ELIGIBILITY:
Inclusion Criteria:

* Require lipid-modifying therapy for primary or secondary prevention of cardiovascular disease
* Fasting LDL-C ≥130 mg/dL for primary prevention or LDL-C ≥100 mg/dL for secondary prevention (history of HeFH and/or ASCVD)
* Be statin-intolerant (unable to tolerate 2 or more statins)

Exclusion Criteria:

* Total fasting triglyceride ≥500 mg/dL
* Renal dysfunction or nephrotic syndrome or history of nephritis
* Body Mass Index (BMI) ≥50 kg/m2
* Significant cardiovascular disease or cardiovascular event in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Haberman, MD, Study Director — Esperion Therapeutics, Inc.
Locations (67):
- United States (52):
  - Gilbert, Arizona
  - Anaheim, California
  - Long Beach, California
  - Sacramento, California
  - Santa Ana, California
  - Torrance, California
  - Ventura, California
  - Hamden, Connecticut
  - Daytona Beach, Florida
  - Fort Lauderdale, Florida
  - Site 1, Miami, Florida
  - Site 2, Miami, Florida
  - Orlando, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Savannah, Georgia
  - Meridian, Idaho
  - Evanston, Illinois
  - Evansville, Indiana
  - Iowa City, Iowa
  - Waterloo, Iowa
  - Monroe, Louisiana
  - Slidell, Louisiana
  - Tupelo, Mississippi
  - Lincoln, Nebraska
  - Somerset, New Jersey
  - Binghamton, New York
  - Endwell, New York
  - New Windsor, New York
  - Greensboro, North Carolina
  - Morganton, North Carolina
  - Mount Airy, North Carolina
  - Columbus, Ohio
  - Marion, Ohio
  - Maumee, Ohio
  - Oklahoma City, Oklahoma
  - Beaver, Pennsylvania
  - Langhorne, Pennsylvania
  - Cumberland, Rhode Island
  - Anderson, South Carolina
  - Summerville, South Carolina
  - Jackson, Tennessee
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Amarillo, Texas
  - Site 1, Dallas, Texas
  - Site 2, Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Clinton, Utah
  - Hampton, Virginia
  - Kenosha, Wisconsin
- Canada (15):
  - Brossard
  - Chicoutimi
  - Gatineau
  - London
  - Longueuil
  - Mirabel
  - Montreal
  - Newmarket
  - Oakville
  - Peterborough
  - Pointe-Claire
  - Saint-Jérôme
  - Sarnia
  - Toronto
  - Victoriaville

REFERENCES:
- [Background] Pinkosky SL, Newton RS, Day EA, Ford RJ, Lhotak S, Austin RC, Birch CM, Smith BK, Filippov S, Groot PHE, Steinberg GR, Lalwani ND. Liver-specific ATP-citrate lyase inhibition by bempedoic acid decreases LDL-C and attenuates atherosclerosis. Nat Commun. 2016 Nov 28;7:13457. doi: 10.1038/ncomms13457. PMID 27892461
- [Background] Cholesterol Treatment Trialists' (CTT) Collaboration; Baigent C, Blackwell L, Emberson J, Holland LE, Reith C, Bhala N, Peto R, Barnes EH, Keech A, Simes J, Collins R. Efficacy and safety of more intensive lowering of LDL cholesterol: a meta-analysis of data from 170,000 participants in 26 randomised trials. Lancet. 2010 Nov 13;376(9753):1670-81. doi: 10.1016/S0140-6736(10)61350-5. Epub 2010 Nov 8. PMID 21067804
- [Background] Eckel RH. Approach to the patient who is intolerant of statin therapy. J Clin Endocrinol Metab. 2010 May;95(5):2015-22. doi: 10.1210/jc.2009-2689. PMID 20444930
- [Background] Ridker PM, Cannon CP, Morrow D, Rifai N, Rose LM, McCabe CH, Pfeffer MA, Braunwald E; Pravastatin or Atorvastatin Evaluation and Infection Therapy-Thrombolysis in Myocardial Infarction 22 (PROVE IT-TIMI 22) Investigators. C-reactive protein levels and outcomes after statin therapy. N Engl J Med. 2005 Jan 6;352(1):20-8. doi: 10.1056/NEJMoa042378. PMID 15635109
- [Background] Robinson JG, Stone NJ. The 2013 ACC/AHA guideline on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular disease risk: a new paradigm supported by more evidence. Eur Heart J. 2015 Aug 14;36(31):2110-2118. doi: 10.1093/eurheartj/ehv182. Epub 2015 May 20. PMID 25994746
- [Derived] Ballantyne CM, Bays HE, Louie MJ, Smart J, Zhang Y, Ray KK. Factors Associated With Enhanced Low-Density Lipoprotein Cholesterol Lowering With Bempedoic Acid. J Am Heart Assoc. 2022 Aug 2;11(15):e024531. doi: 10.1161/JAHA.121.024531. Epub 2022 Aug 2. PMID 35916348
- [Derived] Banach M, Duell PB, Gotto AM Jr, Laufs U, Leiter LA, Mancini GBJ, Ray KK, Flaim J, Ye Z, Catapano AL. Association of Bempedoic Acid Administration With Atherogenic Lipid Levels in Phase 3 Randomized Clinical Trials of Patients With Hypercholesterolemia. JAMA Cardiol. 2020 Oct 1;5(10):1124-1135. doi: 10.1001/jamacardio.2020.2314. PMID 32609313
- [Derived] Laufs U, Banach M, Mancini GBJ, Gaudet D, Bloedon LT, Sterling LR, Kelly S, Stroes ESG. Efficacy and Safety of Bempedoic Acid in Patients With Hypercholesterolemia and Statin Intolerance. J Am Heart Assoc. 2019 Apr 2;8(7):e011662. doi: 10.1161/JAHA.118.011662. PMID 30922146
- See also: World Health Organization Fact Sheet No. 317 — http://www.who.int/mediacentre/factsheets/fs317/en/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 602 participants were screened; out of 602, 345 participants were randomized. 76 participants discontinued investigational medicinal product (IMP), and 18 participants withdrew from the study.
Groups:
- Bempedoic Acid: Participants received a bempedoic acid 180 milligram (mg) tablet taken orally once a day.
- Placebo: Participants received matching oral placebo once a day.
Period: Overall Study
Arm/Group | Bempedoic Acid | Placebo
Started | 234 | 111
Completed | 220 | 107
Not Completed | 14 | 4
Not completed — Adverse Event | 6 | 1
Not completed — Sponsor Decision | 5 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Withdrawn by Mistake | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Bempedoic Acid: Participants received bempedoic acid 180 milligram (mg) tablet taken orally once a day.
- Total: Total of all reporting groups
Arm/Group | Bempedoic Acid | Placebo | Total
Number analyzed (Participants) | 234 | 111 | 345
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.2 (9.66) | 65.1 (9.21) | 65.2 (9.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 61 | 194
  Male | 101 | 50 | 151
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 16 | 10 | 26
  White | 211 | 96 | 307
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Baseline LCL-C, Non-HDL-C, TC, HDL-C, and TG Values [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] — Baseline is defined as the mean of the last two non-missing values on or prior to Day 1. LDL-C, low-density lipoprotein cholesterol; Non-HDL-C, non-high-density lipoprotein cholesterol; TC, total cholesterol; HDL-C, high-density lipoprotein cholesterol; and TG, triglycerides.
  milligrams per deciliter (mg/dL)
    LDL-C | 158.48 (40.387) | 155.58 (38.812) | 157.55 (39.854)
    Non-HDL-C | 193.49 (45.101) | 190.69 (43.781) | 192.59 (44.637)
    TC | 245.66 (47.252) | 241.09 (44.289) | 244.19 (46.304)
    HDL-C | 52.17 (14.535) | 50.41 (14.384) | 51.60 (14.489)
    TG | 178.96 (87.522) | 186.62 (96.203) | 181.42 (90.336)
Baseline Apolipoprotein B (apoB) [Mean (Standard Deviation); unit: mg/dL] — Baseline is defined as the last non-missing value on or prior to Day 1. Population: Only those participants with available data were analyzed.
  mg/dL
    number analyzed (Participants) | 231 | 107 | 338
    (all) | 141.0 (31.64) | 141.9 (30.44) | 141.3 (31.22)
Baseline High-Sensitivity C-Reactive Protein (hsCRP) Values [Median (Full Range); unit: milligrams per liter (mg/L)] — Baseline is defined as the last non-missing value on or prior to Day 1. Population: Only those participants with available data were analyzed.
  milligrams per liter (mg/L)
    number analyzed (Participants) | 231 | 106 | 337
    (all) | 2.920 [1.340 to 5.290] | 2.780 [1.210 to 5.150] | 2.900 [1.290 to 5.150]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline (PCFB) in Low-density Lipoprotein Cholesterol (LDL-C) at Week 12
Description: PCFB was calculated as the ([post-Baseline (BL) value minus the BL value] divided by the BL value ) x 100. BL was defined as the mean of the last two non-missing values on or prior to Day 1. If only one value was available, that single value was used as BL. PCFB in LDL-C was analyzed using analysis of covariance (ANCOVA), with treatment group and stratification factor (primary prevention; secondary prevention) as fixed effects and BL as a covariate. For participants with missing lipid data at Week 12 who were no longer taking study treatment, missing values were imputed using multiple imputation via a regression-based model including stratification and BL data from placebo participants only. In this imputation model, treatment group was not included. For participants with missing lipid data at Week 12 who were still taking study treatment, missing values were imputed using multiple imputation via a regression-based model including treatment, stratification and BL value.
Time Frame: Baseline; Week 12
Population: The Full Analysis Set (FAS), also known as the intention-to-treat (ITT) set of participants, is defined as all randomized participants. Participants were included in their randomized treatment group, regardless of the treatment they actually received. Only those participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Bempedoic Acid | Placebo
Number analyzed (Participants) | 224 | 107
percent change | -22.58 (1.290) | -1.17 (1.421)
Statistical Analysis 1: Comparison: Bempedoic Acid vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; Least squares means difference = -21.41, 95% CI 2-sided [-25.132 to -17.697], Standard Error of Mean 1.897 — bempedoic acid (BA) therapy minus placebo

2. Secondary Outcome: Percent Change From Baseline in LDL-C at Week 24
Description: PCFB was calculated as the ([post-BL value minus the BL value] divided by the BL value ) x 100. BL was defined as the mean of the last two non-missing values on or prior to Day 1. If only one value was available then that single value was used as BL. PCFB in LDL-C was analyzed using ANCOVA, with treatment group and stratification factor (primary prevention; secondary prevention) as fixed effects and BL as a covariate. For participants with missing lipid data at Week 12 who were no longer taking study treatment, missing values were imputed using multiple imputation via a regression-based model including stratification and BL data from placebo participants only. In this imputation model, treatment group was not included. For participants with missing lipid data at Week 12 who were still taking study treatment, missing values were imputed using multiple imputation via a regression-based model including treatment, stratification and BL value.
Time Frame: Baseline; Week 24
Population: FAS. Only those participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Bempedoic Acid | Placebo
Number analyzed (Participants) | 217 | 106
percent change | -21.17 (1.411) | -2.26 (1.552)
Statistical Analysis 1: Comparison: Bempedoic Acid vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; Least squares means difference = -18.91, 95% CI 2-sided [-22.951 to -14.865], Standard Error of Mean 2.063 — BA therapy minus placebo

3. Secondary Outcome: Percent Change From Baseline in the Lipid Profile at Week 12
Description: PCFB was calculated as: ([post-BL value minus the BL value] divided by the BL value) x 100. BL was defined as the mean of the last two non-missing values on or prior to Day 1. If only one value was available, that single value was used as BL. apoB and TC BL were defined as the last non-missing value on/prior to Day 1. PCFB was analyzed using ANCOVA, with treatment and group stratification factor (primary prevention; secondary prevention) as fixed effects and BL as a covariate. For participants with missing data at Week 12 who were no longer taking study treatment (ST), missing values were imputed using multiple imputation via a regression-based model including stratification and BL data from placebo participants only. In this imputation model, treatment group was not included. For participants with missing lipid data at Week 12 who were still taking ST, missing values were imputed using multiple imputation via a regression-based model including treatment, stratification and BL value.
Time Frame: Baseline; Week 12
Population: FAS. Only those participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Bempedoic Acid | Placebo
Number analyzed (Participants) | 224 | 107
percent change
  non-HDL-C | -18.08 (1.114) | -0.14 (1.169)
  TC | -15.37 (0.879) | -0.61 (0.961)
  apoB: number analyzed (Participants) | 218 | 104
  apoB | -14.65 (1.080) | 0.32 (1.177)
Statistical Analysis 1: Comparison: Bempedoic Acid vs Placebo; non-HDL-C; Test type: Superiority; p < 0.001, ANCOVA; Least squares means difference = -17.94, 95% CI 2-sided [-21.070 to -14.811], Standard Error of Mean 1.597 — BA therapy minus placebo
Statistical Analysis 2: Comparison: Bempedoic Acid vs Placebo; TC; Test type: Superiority; p < 0.001, ANCOVA; Least squares means difference = -14.76, 95% CI 2-sided [-17.283 to -12.239], Standard Error of Mean 1.287 — BA therapy minus placebo
Statistical Analysis 3: Comparison: Bempedoic Acid vs Placebo; apoB; Test type: Superiority; p < 0.001, ANCOVA; Least squares means difference = -14.96, 95% CI 2-sided [-18.062 to -11.866], Standard Error of Mean 1.581 — BA therapy minus placebo

4. Secondary Outcome: Percent Change From Baseline in High-Sensitivity C-Reactive Protein (hsCRP) at Week 12
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline for hsCRP is defined as the last non-missing value on or prior to Day 1. Percent change from Baseline in hsCRP, non-parametric (Wilcoxon rank-sum test) analysis with Hodges-Lehmann estimates and confidence interval was performed.
Time Frame: Baseline; Week 12
Population: FAS. Only those participants with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Bempedoic Acid | Placebo
Number analyzed (Participants) | 218 | 103
percent change | -25.37 [-52.75 to 10.78] | 2.67 [-31.07 to 38.04]
Statistical Analysis 1: Comparison: Bempedoic Acid vs Placebo; Test type: Superiority; p < 0.001, Wilcoxon rank sum test; Median treatment difference = -24.290, 95% CI 2-sided [-35.888 to -12.712], Standard Error of Mean -24.300 — BA therapy minus placebo

5. Secondary Outcome: Absolute Change From Baseline in LDL-C at Week 12 and Week 24
Description: Change from Baseline is calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value ) x 100. Baseline is defined as the mean of the last two non-missing values on or prior to Day 1.
Time Frame: Baseline; Week 12; Week 24
Population: FAS. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Bempedoic Acid | Placebo
Number analyzed (Participants) | 224 | 107
mg/dL
  Week 12 | -39.3 (33.37) | -3.1 (23.66)
  Week 24: number analyzed (Participants) | 217 | 106
  Week 24 | -37.0 (35.27) | -5.1 (26.50)

ADVERSE EVENTS:
Time Frame: Up to 24 weeks plus 30 days
Description: Treatment-emergent adverse events (TEAEs), defined as those events that began or worsened after the first dose of IMP until 30 days after the last dose of IMP, were reported for the Safety Population. The Safety Population is defined as all randomized participants who received at least 1 dose of double-blind study medication.
Arm/Group | Bempedoic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/234 | 0/111
Serious Adverse Events (participants affected / at risk) | 14/234 | 4/111
Other Adverse Events (participants affected / at risk) | 88/234 | 45/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bempedoic Acid (N=234) | Placebo (N=111)
Angina unstable (Cardiac disorders) | 3 | 0
Coronary artery disease (Cardiac disorders) | 3 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Cerebrovascular accident (Blood and lymphatic system disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Corneal lesion (Eye disorders) | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0
Ischaemic stroke (Blood and lymphatic system disorders) | 1 | 0
Lower respiratory tract infection bacterial (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Myeloproliferative neoplasm (Blood and lymphatic system disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Staphylococcal infection (Skin and subcutaneous tissue disorders) | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Aortic aneurysm (Cardiac disorders) | 0 | 1
Escherichia pyelonephritis (Renal and urinary disorders) | 0 | 1
Escherichia sepsis (Blood and lymphatic system disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Traumatic intracranial haemorrhage (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bempedoic Acid (N=234) | Placebo (N=111)
Dyspepsia (Gastrointestinal disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 4 | 3
Fatigue (General disorders) | 8 | 7
Bronchitis (Infections and infestations) | 6 | 6
Nasopharyngitis (Infections and infestations) | 3 | 5
Upper respiratory tract infection (Infections and infestations) | 2 | 3
Urinary tract infection (Infections and infestations) | 7 | 9
Blood creatine phosphokinase increased (Investigations) | 5 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 8
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 4
Dizziness (Nervous system disorders) | 7 | 0
Headache (Nervous system disorders) | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Hypertension (Vascular disorders) | 10 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the Principal Investigator plans to publish information from the study, a copy of the manuscript should be provided to the Sponsor for review before submission for publication or presentation. The Sponsor may request that publication be withheld.

DOCUMENTS (2):
  • Study Protocol (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT02988115/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/15/NCT02988115/SAP_001.pdf